CLINICAL TRIAL: NCT05186298
Title: Prospective Evaluation and Comparison of Bilateral Synergy Implants and Bilateral PanOptix Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alterman, Modi, & Wolter Ophthalmic Physicians & Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 68985013
Record Dates: First submitted 2021-11-16; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- AcrySof® IQ PanOptix® (Alcon Laboratories, Inc., Fort Worth, TX) (Experimental): The subject will be implanted bilaterally during cataract surgery
  Interventions: Device: AcrySof® IQ PanOptix®; Procedure: Cataract Surgery
- Synergy® (Johnson & Johnson Surgical Vision, Santa Ana, CA) (Experimental): The subject will be implanted bilaterally during cataract surgery
  Interventions: Device: Synergy®; Procedure: Cataract Surgery

INTERVENTIONS:
Device: AcrySof® IQ PanOptix® — The AcrySof IQ PanOptix® (Alcon) mitigates the effects of presbyopia by providing improved intermediate and near visual acuity, while maintaining comparable distance visual acuity with a reduced need for eyeglasses, compared to a monofocal IOL
  Arms: AcrySof® IQ PanOptix® (Alcon Laboratories, Inc., Fort Worth, TX)
Device: Synergy® — The TECNIS Synergy™ IOLs mitigate the effects of presbyopia by providing far vision comparable to an aspheric monofocal IOL. Compared to an aspheric monofocal IOL, the lens provides significantly improved intermediate and near vision, including in low-light conditions.
  Arms: Synergy® (Johnson & Johnson Surgical Vision, Santa Ana, CA)
Procedure: Cataract Surgery — IOL implantation will be performed

SUMMARY:
The purpose of this study is to evaluate the AcrySof PanOptix Intraocular Lens (IOL) for binocular distance corrected near visual acuity (DCNVA) compared to TECNIS Synergy IOL.

Presbyopia correcting diffractive intraocular implants (extended depth of focus, multifocal, and trifocal) provide cataract and refractive surgeons with an effective treatment means for allowing patients to experience increased spectacle independence post-cataract surgery.

DETAILED DESCRIPTION:
Eligible test subjects will be patients diagnosed with cataracts bilaterally who are interested and eligible for implantation of a presbyopia-correcting multifocal intraocular lenses.

Subjects will participate in ten study visits. Visits will include a screening visit (both eyes evaluated), one operative visit for each eye, and 7 postoperative visits. Both eyes will be implanted, with the second eye surgery occurring X (depends on the patient and the schedule) days after the first.

ELIGIBILITY:
Inclusion Criteria:

Note: Ocular criteria must be met in both eyes.

* are willing and able to understand and sign an informed consent;
* are willing and able to attend all study visits;
* Subjects diagnosed with bilateral cataracts with planned cataract removal by femto assisted phacoemulsification with a clear corneal incision and intraoperative aberrometry assisted
* Clear intraocular media other than cataracts.
* Projected BCDVA of better than 0.10 logMAR.
* Preoperative regular keratometric astigmatism (by biometer) of less than or equal to 0.75D, in both eyes
* Biometer IOL calculations within +6.0 - +30.0 power range

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Clinically significant corneal abnormality, irregularity, inflammation, or edema aberrations, corneal disease, degeneration, or conditions affecting postoperative visual acuity
* Glaucoma or Ocular Hypertension
* Planned multiple procedures (eg MIGS)
* Amblyopia, Strabismus
* Patient's IOL calculation that are outside the range of available lenses
* Prior corneal refractive surgery or other corneal surgery (e.g., corneal transplant, lamellar keratoplasty, LASIK, PRK)
* Previous anterior or posterior chamber surgery (e.g., vitrectomy) that the investigator feels may compromise visual outcomes
* Diabetic retinopathy if the investigator feels this will compromise visual outcomes
* Macular Pathology (i.e., ERM, ARMD, DMR etc.) if the investigator feels this will compromise visual outcomes
* History of retinal detachment
* If, in the surgeon's opinion, the subject is not an appropriate candidate for multifocal IOL implantation (eg. patients who are professional night drivers or pilots, and those with other occupations for whom induces dysphotopsias could put their career at risk)
* Subjects who have an acute or chronic disease or illness that would confound the results of this investigation (e.g., immunocompromised, connective tissue disease, clinically significant atopic disease, diabetes, and any other such disease or illness), that are known to affect post-operative visual acuity.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Binocular DCNVA | Up to Month 6
  Binocular DCNVA of Trifocal (Alcon Panoptix) versus EDOF/Bifocal (Johnson and Johnson Tecnis Synergy) at 40 cm

SECONDARY OUTCOMES:
Visual Disturbances Evaluation | at all visits
  Patient reported occurrences of visual disturbances of each group (unsolicited) at all visits
Visual Disturbances Evaluation by Questionnaire (QUVID) | Up to Month 6
  Patient reported visual disturbances by questionnaire (QUVID) postop
BCDVA and DCIVA (60 cm) | Up to Month 6
  Monocular and binocular BCDVA and DCIVA (60 cm) in both groups will be measured
DCNVA (40 cm) | Up to Month 6
  Monocular DCNVA (40 cm) in both groups will be measured
Uncorrected Monocular and Binocular VA | Up to Month 6
  Uncorrected monocular and binocular VA at distance, intermediate (60 cm) and near (40 cm)
Visual Disturbances Evaluation by Questionnaire (IOL SAT) | Up to Month 6
  Patient satisfaction of each group by questionnaire (IOL SAT) postop
Defocus Curve | Up to Month 6
  Defocus curve tested in binocular photopic conditions (+1.00 to -3.00 in 0.50D except +0.50 to -0.50 in 0.25D)

CONTACTS AND LOCATIONS:
Overall Officials: Satish S Modi, MD, Principal Investigator — Seeta Eye Centre
Locations (5):
- United States (5):
  - Eye Care Now, Panama City, Florida
  - Seeta Eye Center, Poughkeepsie, New York
  - Eye Care Specialists, Kingston, Pennsylvania
  - Lehmann Eye Center, Nacogdoches, Texas
  - Northwest Eye Surgeons, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Modi SS, Lehmann RP, Fisher BL, Roth RE, Reiser H. Comparison of visual function and patient-reported outcomes between two full range of field intraocular lenses: a randomized controlled study. J Cataract Refract Surg. 2025 Aug 1;51(8):695-702. doi: 10.1097/j.jcrs.0000000000001678. PMID 40277405